CLINICAL TRIAL: NCT03226886
Title: TRACERx Renal (TRAcking Renal Cell Carcinoma Evolution Through Therapy (Rx)) CAPTURE: COVID-19 Antiviral Response in a Pan-tumour Immune Study
Brief Title: TRACERx Renal CAPTURE Sub-study
Acronym: TRACERxRenal
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Francis Crick Institute (Other)
Responsible Party: Sponsor
Other Study IDs: CCR 3723
Record Dates: First submitted 2017-07-06; First posted 2017-07-24 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2019-09

CONDITIONS: Renal Cell Carcinoma; Cancer; Healthy Volunteers
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — TRACERx Renal: The Investigators will be collecting Blood, Urine, Core Biopsies and Surgical Samples
  CAPTURE Sub-study: The Investigators will be collecting Bloods, Swabs and stored samples from patients and Health Care Workers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients: In London renal cell carcinoma patients undergo nephrectomy at centres for urological oncology, including the Royal Marsden, Guy's and St Thomas', St Georges, Charing Cross and Kings Hospitals. It is not uncommon for the same patients to undergo palliative resection for metastatic sites of disease. The majority of tissue from these resections does not undergo routine histopathological examination. As such, it is ethically feasible to use these specimens for laboratory research in the presence of patient consent. Practically, these specimens are often large, thereby offering considerable scope for a range of molecular analyses.
  CAPTURE Sub-study:
  We plan to enrol patients/participants into three groups:
  Group A: patients with confirmed or suspected COVID-19 and a history of cancer Group B: patients without a history of COVID-19 infection and a history of cancer Group C: Hospital staff with or without a history of COVID-19

SUMMARY:
TRACERx Renal: This is a translational study, which, aims to develop prognostic and predictive biomarkers for patients with renal cell carcinoma (RCC).

CAPTURE Sub-study: Covid-19 antiviral response in a pan-tumour immune monitoring study

DETAILED DESCRIPTION:
There is a need for improved understanding of renal cell carcinoma (RCC) biology in order to characterise the mechanisms of metastatic progression, drug resistance, develop predictive & prognostic biomarkers and to identify novel therapeutic targets for this disease. The TRACERx consortium was established to achieve this using large longitudinal clinical studies, in collaboration with laboratory, advanced sequencing and informatics expertise to identify the relationships between intratumour heterogeneity and clinical outcome.

Response and Resistance: TRACERx Renal is a prospective longitudinal cohort study. It will draw on the methodology already being used within the TRACERx Lung & (planned) Breast studies as part of the TRACERx consortium.

Primary Endpoint

• To validate ITH index and WGII as stage and grade independent prognostic markers of progression free survival in patients with ccRCC

The Investigators plan to collect the following biological samples:

* Blood sample/s, urine and tumour biopsy tissue taken prior to any neoadjuvant treatment that might be administered.
* Blood sample/s, urine and tumour biopsy tissue taken prior to any ablative procedure
* Blood sample/s, urine and nephrectomy tissue taken at the time of nephrectomy.
* Blood sample/s, urine and tumour tissue taken at the time of palliative metastasectomy/surgery.
* Blood and urine sample/s taken at routine follow up.
* Blood sample/s, urine and tumour biopsy taken at time of disease progression.
* Blood sample/s and/or archival tissue specimens that are no longer required by the local pathologist for diagnostic purposes
* Blood sample/s and/or archival tissue specimens that are no longer required by the local pathologist for diagnostic purposes from study patient family members

CAPTURE sub-study:

There is an urgent need to quantify the risk of COVID-19 illness in patients with cancer and to understand what impact anti-cancer treatments have on the immune system's response to the SARS-CoV-2 virus. There is also a need to understand how the pandemic impacts Health Care Workers (HCWs) who may be exposed to the virus in the course of their clinical duties and who are at risk to transmit the virus to vulnerable patients and colleagues in the asymptomatic phase of infection.

The CAPTURE study is a long-term study. We are establishing large observational cohorts with an intentionally broad inclusion of different tumour types and treatment schedules. In CAPTURE, we will enrol both patients infected and uninfected by the virus, and patients with all types of cancer (blood and solid cancers), and of all walks of the clinical journey (in remission, follow-up, having treatment or undergoing surgery). We also will enrol HCWs within the hospital from all sectors of care delivery - from nurses to doctors, administrative staff to catering staff, allied health and support workers.

The study will enrol patients/participants into three groups:

Group A: patients with confirmed or suspected COVID-19 and a history of cancer (n=200) Group B: patients without a history of COVID-19 infection and a history of cancer (n=1000) Group C: Hospital staff with or without a history of COVID-19 (n=200)

Comprehensive, longitudinal clinical annotation, participant questionnaires, meticulous and frequent sampling and long-term follow-up of these groups will allow robust and rapid insights that are urgently needed to guide clinical and workforce management.

This knowledge is required well beyond the current pandemic as cancer and SARSCo-V2 will coincide in the same patients, and especially given the uncertainty regarding the nature and duration of immunity in cancer patients who develop the illness and the effectiveness of vaccines in the cancer population. This study will provide us with detailed information on how to safely manage cancer patients by both minimising the risk of infection but maintaining their cancer treatment.

ELIGIBILITY:
TRACERx Renal Inclusion Criteria:

* Age 18- years or older
* Patients with histopathologically confirmed renal cell carcinoma, or suspected renal cell carcinoma, proceeding to neoadjuvant therapy and/or nephrectomy/metastasectomy, or identified as having progressive disease
* Or in patients undergoing nephrectomy for non-malignant disease
* Medical and/or surgical management in accordance with national and/or local guidelines
* Written informed consent

Exclusion Criteria:

* Any concomitant medical or psychiatric problems which, in the opinion of the investigator, would prevent completion of treatment or follow-up
* Lack of adequate tissue

CAPTURE Inclusion criteria

* Documented informed consent
* Age 18 years or older
* Confirmed cancer diagnosis (irrespective of cancer type, disease burden or treatment)
* Group A: Suspected infection with SARS-CoV-2 or positive test for SARS-CoV-2
* Group B: no clinical indication to test for SARS-CoV-2 (by current Trust guidelines*) or tested negative for SARS-CoV-2
* Group C: Volunteers without cancer with SARS-CoV-2 (symptomatic and asymptomatic) and those without clinical indication (current national guidelines*) for SARS-CoV-2 testing or tested negative for SARS-CoV-2

Exclusion criteria

• Medical or psychological condition that would preclude informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: TRACERx Renal: Patients with histopathologically confirmed renal cell carcinoma, or suspected renal cell carcinoma, proceeding to neoadjuvant therapy and/or nephrectomy/metastectomy, or identified as having progressive disease or in patients undergoing nephrectomy for non-malignant disease
  CAPTURE:
  Group A : Cancer patients with SARS-CoV-2 Group B : Cancer patients without clinical indication for SARS-CoV-2 testing (based on current local guidelines) or have tested negative for SARS-CoV-2 Group C: Volunteers without cancer (recruiting site staff)
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2012-02-05 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
To validate ITH index and WGII as stage and grade independent prognostic markers of progression free survival in patients with ccRCC mutation in a gene of interest | From trial activation until trial closure approximately 1st September 2023
  Outcomes will be quantified using descriptive statistics with the intention of providing hypothesis-generating data for use in future studies.
CAPTURE Sub-study: Describe the population characteristics between SARS-CoV-2 positive and negative cancer patients | From sub-study activation until trial closure approximately 2027
  Outcomes will be quantified using descriptive statistics

CONTACTS AND LOCATIONS:
Overall Officials: Samra Turajlic, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (4):
- United Kingdom (4):
  - Edinburgh Western General Hospital, Edinburgh, Scotland
  - Guy's & St Thomas Hospital, London, UK
  - Barts Health NHS Trust, London
  - Royal Free Hospital, London

IPD SHARING:
Plan to Share IPD: No
Patients are given a unique identifier as soon as they are consented. All samples and data is anonymised and can only be accessed by the research team.

REFERENCES:
- [Derived] Orton MR, Hann E, Doran SJ, Shepherd STC, Ap Dafydd D, Spencer CE, Lopez JI, Albarran-Artahona V, Comito F, Warren H, Shur J, Messiou C, Larkin J, Turajlic S; TRACERx Renal Consortium; Koh DM. Interpretability of radiomics models is improved when using feature group selection strategies for predicting molecular and clinical targets in clear-cell renal cell carcinoma: insights from the TRACERx Renal study. Cancer Imaging. 2023 Aug 14;23(1):76. doi: 10.1186/s40644-023-00594-3. PMID 37580840
- [Derived] Piening A, Ebert E, Khojandi N, Alspach E, Teague RM. Immune responses to SARS-CoV-2 in vaccinated patients receiving checkpoint blockade immunotherapy for cancer. Front Immunol. 2022 Dec 13;13:1022732. doi: 10.3389/fimmu.2022.1022732. eCollection 2022. PMID 36582225
- [Derived] Fendler A, Shepherd STC, Au L, Wu M, Harvey R, Wilkinson KA, Schmitt AM, Tippu Z, Shum B, Farag S, Rogiers A, Carlyle E, Edmonds K, Del Rosario L, Lingard K, Mangwende M, Holt L, Ahmod H, Korteweg J, Foley T, Barber T, Emslie-Henry A, Caulfield-Lynch N, Byrne F, Deng D, Kjaer S, Song OR, Queval CJ, Kavanagh C, Wall EC, Carr EJ, Caidan S, Gavrielides M, MacRae JI, Kelly G, Peat K, Kelly D, Murra A, Kelly K, O'Flaherty M, Shea RL, Gardner G, Murray D, Popat S, Yousaf N, Jhanji S, Tatham K, Cunningham D, Van As N, Young K, Furness AJS, Pickering L, Beale R, Swanton C, Gandhi S, Gamblin S, Bauer DLV, Kassiotis G, Howell M, Nicholson E, Walker S, Wilkinson RJ, Larkin J, Turajlic S. Functional immune responses against SARS-CoV-2 variants of concern after fourth COVID-19 vaccine dose or infection in patients with blood cancer. Cell Rep Med. 2022 Oct 18;3(10):100781. doi: 10.1016/j.xcrm.2022.100781. Epub 2022 Sep 27. PMID 36240755
- [Derived] Fendler A, Shepherd STC, Au L, Wilkinson KA, Wu M, Byrne F, Cerrone M, Schmitt AM, Joharatnam-Hogan N, Shum B, Tippu Z, Rzeniewicz K, Boos LA, Harvey R, Carlyle E, Edmonds K, Del Rosario L, Sarker S, Lingard K, Mangwende M, Holt L, Ahmod H, Korteweg J, Foley T, Bazin J, Gordon W, Barber T, Emslie-Henry A, Xie W, Gerard CL, Deng D, Wall EC, Agua-Doce A, Namjou S, Caidan S, Gavrielides M, MacRae JI, Kelly G, Peat K, Kelly D, Murra A, Kelly K, O'Flaherty M, Dowdie L, Ash N, Gronthoud F, Shea RL, Gardner G, Murray D, Kinnaird F, Cui W, Pascual J, Rodney S, Mencel J, Curtis O, Stephenson C, Robinson A, Oza B, Farag S, Leslie I, Rogiers A, Iyengar S, Ethell M, Messiou C, Cunningham D, Chau I, Starling N, Turner N, Welsh L, van As N, Jones RL, Droney J, Banerjee S, Tatham KC, O'Brien M, Harrington K, Bhide S, Okines A, Reid A, Young K, Furness AJS, Pickering L, Swanton C; Crick COVID-19 Consortium; Gandhi S, Gamblin S, Bauer DLV, Kassiotis G, Kumar S, Yousaf N, Jhanji S, Nicholson E, Howell M, Walker S, Wilkinson RJ, Larkin J, Turajlic S; CAPTURE Consortium. Adaptive immunity and neutralizing antibodies against SARS-CoV-2 variants of concern following vaccination in patients with cancer: the CAPTURE study. Nat Cancer. 2021 Dec;2(12):1305-1320. doi: 10.1038/s43018-021-00274-w. Epub 2021 Oct 27. PMID 35121899
- [Derived] Fendler A, Shepherd STC, Au L, Wilkinson KA, Wu M, Byrne F, Cerrone M, Schmitt AM, Joharatnam-Hogan N, Shum B, Tippu Z, Rzeniewicz K, Boos LA, Harvey R, Carlyle E, Edmonds K, Del Rosario L, Sarker S, Lingard K, Mangwende M, Holt L, Ahmod H, Korteweg J, Foley T, Bazin J, Gordon W, Barber T, Emslie-Henry A, Xie W, Gerard CL, Deng D, Wall EC, Agua-Doce A, Namjou S, Caidan S, Gavrielides M, MacRae JI, Kelly G, Peat K, Kelly D, Murra A, Kelly K, O'Flaherty M, Dowdie L, Ash N, Gronthoud F, Shea RL, Gardner G, Murray D, Kinnaird F, Cui W, Pascual J, Rodney S, Mencel J, Curtis O, Stephenson C, Robinson A, Oza B, Farag S, Leslie I, Rogiers A, Iyengar S, Ethell M, Messiou C, Cunningham D, Chau I, Starling N, Turner N, Welsh L, van As N, Jones RL, Droney J, Banerjee S, Tatham KC, O'Brien M, Harrington K, Bhide S, Okines A, Reid A, Young K, Furness AJS, Pickering L, Swanton C; Crick COVID19 consortium; Gandhi S, Gamblin S, Bauer DL, Kassiotis G, Kumar S, Yousaf N, Jhanji S, Nicholson E, Howell M, Walker S, Wilkinson RJ, Larkin J, Turajlic S. Adaptive immunity and neutralizing antibodies against SARS-CoV-2 variants of concern following vaccination in patients with cancer: The CAPTURE study. Nat Cancer. 2021 Dec;2:1321-1337. doi: 10.1038/s43018-021-00274-w. Epub 2021 Oct 27. PMID 34950880
- [Derived] Turajlic S, Xu H, Litchfield K, Rowan A, Chambers T, Lopez JI, Nicol D, O'Brien T, Larkin J, Horswell S, Stares M, Au L, Jamal-Hanjani M, Challacombe B, Chandra A, Hazell S, Eichler-Jonsson C, Soultati A, Chowdhury S, Rudman S, Lynch J, Fernando A, Stamp G, Nye E, Jabbar F, Spain L, Lall S, Guarch R, Falzon M, Proctor I, Pickering L, Gore M, Watkins TBK, Ward S, Stewart A, DiNatale R, Becerra MF, Reznik E, Hsieh JJ, Richmond TA, Mayhew GF, Hill SM, McNally CD, Jones C, Rosenbaum H, Stanislaw S, Burgess DL, Alexander NR, Swanton C; PEACE; TRACERx Renal Consortium. Tracking Cancer Evolution Reveals Constrained Routes to Metastases: TRACERx Renal. Cell. 2018 Apr 19;173(3):581-594.e12. doi: 10.1016/j.cell.2018.03.057. Epub 2018 Apr 12. PMID 29656895
- [Derived] Turajlic S, Xu H, Litchfield K, Rowan A, Horswell S, Chambers T, O'Brien T, Lopez JI, Watkins TBK, Nicol D, Stares M, Challacombe B, Hazell S, Chandra A, Mitchell TJ, Au L, Eichler-Jonsson C, Jabbar F, Soultati A, Chowdhury S, Rudman S, Lynch J, Fernando A, Stamp G, Nye E, Stewart A, Xing W, Smith JC, Escudero M, Huffman A, Matthews N, Elgar G, Phillimore B, Costa M, Begum S, Ward S, Salm M, Boeing S, Fisher R, Spain L, Navas C, Gronroos E, Hobor S, Sharma S, Aurangzeb I, Lall S, Polson A, Varia M, Horsfield C, Fotiadis N, Pickering L, Schwarz RF, Silva B, Herrero J, Luscombe NM, Jamal-Hanjani M, Rosenthal R, Birkbak NJ, Wilson GA, Pipek O, Ribli D, Krzystanek M, Csabai I, Szallasi Z, Gore M, McGranahan N, Van Loo P, Campbell P, Larkin J, Swanton C; TRACERx Renal Consortium. Deterministic Evolutionary Trajectories Influence Primary Tumor Growth: TRACERx Renal. Cell. 2018 Apr 19;173(3):595-610.e11. doi: 10.1016/j.cell.2018.03.043. Epub 2018 Apr 12. PMID 29656894
- See also: TRACERx Consortium Website — http://tracerx.co.uk/studies/renal/